CLINICAL TRIAL: NCT03002831
Title: Autologous Cytokine-induced Killer Cells Combined Chemotherapy in Advanced Pancreatic Cancer: A Prospective, Randomized, Open, Single Center Phase II Study
Brief Title: Autologous Cytokine-induced Killer Cells Combined Chemotherapy in Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH CIK02
Record Dates: First submitted 2016-12-19; First posted 2016-12-26 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2016-12

CONDITIONS: Advanced Cancer
Keywords: CIK; Chemotherapy; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIK combined chemotherapy (Experimental): Autologous Cytokine induced killer cells combined Tegafur, Gimeracil and Oteracil Potassium Capsules. After 2 to 4 days of chemotherapy, about 5×10９autologous cytokine induced killer cells are transfused into the vein of the patients in one hour.
  Interventions: Biological: Cytokine-induced Killer Cells; Drug: Tegafur-Gimeracil-Oteracil Potassium
- Chemotherapy (Active Comparator): Tegafur,Gimeracil and Oteracil Potassium Capsules 40-60mg, bid, po, D1-14, Q3w
  Interventions: Drug: Tegafur-Gimeracil-Oteracil Potassium

INTERVENTIONS:
Biological: Cytokine-induced Killer Cells
  Arms: CIK combined chemotherapy
Drug: Tegafur-Gimeracil-Oteracil Potassium

SUMMARY:
The purpose of this study is to determine whether Cytokine induced killer cells combined chemotherapy is more effective in the treatment of advanced Pancreatic Cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is a devastating malignant disease with a median survival of 3-6 months and a 5-year survival rate of less than 5%. It is necessary to explore more treatment mode to pancreatic cancer especially advanced stage patients. This study is a prospective, randomized, open, single center phase II study. The investigators try to evaluate the efficacy and safety of this treatment mode.

ELIGIBILITY:
Inclusion Criteria:

1. No less than 18 years old
2. Karnofsky Performance Status over 60
3. Life expectancy more than three months
4. Pathological diagnosed as pancreatic epithelial cell carcinoma
5. Recurrence after surgery or unresectable
6. No experienced chemotherapy or the interval between the last adjuvant chemotherapy and relapse is at least 6 months
7. Measurable lesions (by CT or MRI)
8. No serious mental disorders
9. Adequate organ and bone marrow functions
10. No other serious and the conflict diseases(such as autoimmune diseases, immunodeficiency, organ transplantation)
11. No other malignant tumor history
12. Informed consent and willing to participate in this study

Exclusion Criteria:

1. Received immunosuppressants or glucocorticoid treatment
2. Uncontrolled severe infection or unhealed wound caused by suppurative inflammation
3. Heart disease, insufficient heart function, II degree heart block or occurred myocardial infarction in 6 months
4. Poor pulmonary functions caused by interstitial lung disease and pulmonary reserve volume under 80% of the expected value
5. Other malignant tumor history
6. Transaminase>2.5ULN or bilirubin>3ULN or creatinine >1.25ULN
7. Pregnant or lactating women
8. Obvious bleeding tendency
9. Participated other clinical trails in 1 month
10. Other unsuitable conditions: HIV infection, intravenous drug abusers, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From the date of randomization to the date of death from any cause up to 36 months

SECONDARY OUTCOMES:
Progression Free Survival | From the date of randomization to the date of first documented progression up to 24 months
Quality of life assessed by Questionnaire | one year by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Quanli Gao, Ph.D., Principal Investigator — Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Imaoka H, Kou T, Tanaka M, Egawa S, Mizuno N, Hijioka S, Hara K, Yazumi S, Shimizu Y, Yamao K. Clinical outcome of elderly patients with unresectable pancreatic cancer treated with gemcitabine plus S-1, S-1 alone, or gemcitabine alone: Subgroup analysis of a randomised phase III trial, GEST study. Eur J Cancer. 2016 Feb;54:96-103. doi: 10.1016/j.ejca.2015.11.002. Epub 2015 Dec 30. PMID 26741729
- [Result] Wang Z, Liu Y, Li R, Shang Y, Zhang Y, Zhao L, Li W, Yang Y, Zhang X, Yang T, Nie C, Han F, Liu Y, Luo S, Gao Q, Song Y. Autologous cytokine-induced killer cell transfusion increases overall survival in advanced pancreatic cancer. J Hematol Oncol. 2016 Feb 3;9:6. doi: 10.1186/s13045-016-0237-6. PMID 26842696